CLINICAL TRIAL: NCT05929573
Title: Efficacy of Renal Doppler Resistive Index and Neutrophil Gelatinase-Associated Lipocalin Measurement in Detecting Acute Kidney Injury in Major Abdominal Surgery
Brief Title: RDRI and NGAL in Acute Kidney Injury in Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erhan Ozyurt, Associate Professor, M.D., Antalya Training and Research Hospital
Other Study IDs: Ercan01
Record Dates: First submitted 2023-06-25; First posted 2023-07-03 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Neutrophil Gelatinase-Associated Lipocalin; Renal Doppler Resistive Index; Major Abdominal Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neutrophil Gelatinase-Associated Lipocalin — Neutrophil Gelatinase-Associated Lipocalin, which can be measured from serum or urine, can detect acute kidney failure that may occur after surgery in the early stages.
Diagnostic Test: Renal Doppler Resistive Index — Renal Doppler Resistive Index (RDRI) is a non-invasive index believed to reflect renal vascular perfusion. RDRI measurement is a repeatable, inexpensive, and easy-to-apply technique. RDRI has been found to be associated with AKI in conditions such as renal dysfunction, hypertension, and post-traumatic hemorrhagic shock. Furthermore, due to the impact on renal perfusion in patients undergoing major surgery, RDRI, which reflects renal vascular resistance, can serve as an indicator of kidney perfusion.

SUMMARY:
Acute kidney injury (AKI), which can occur after major surgeries, leads to increased morbidity and mortality if not detected and managed promptly. In clinical practice, serum creatinine and urine output values of patients are monitored to detect AKI, but these parameters can cause delays in diagnosis. Additionally, studies have been conducted on biomarkers such as Neutrophil Gelatinase-Associated Lipocalin (NGAL) and cystatin C in recent years, but definitive results have not been achieved.

Renal Doppler Resistive Index (RDRI) is a non-invasive index believed to reflect renal vascular perfusion. RDRI measurement is a repeatable, inexpensive, and easy-to-apply technique. RDRI has been found to be associated with AKI in conditions such as renal dysfunction, hypertension, and post-traumatic hemorrhagic shock. Furthermore, due to the impact on renal perfusion in patients undergoing major surgery, RDRI, which reflects renal vascular resistance, can serve as an indicator of kidney perfusion.

The aim of this study is to test the hypothesis, 'Does measuring postoperative RDRI in major abdominal surgery cases yield higher sensitivity and specificity values in detecting acute kidney injury compared to NGAL?'

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III,
* Patients undergoing elective major abdominal surgery

Exclusion Criteria:

* Chronic kidney failure,
* Using nephrotoxic drugs,
* Patients with a history of kidney transplantation or nephrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo major abdominal surgery in Antalya Training and Research Hospital.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Plasma NGAL Level | Postoperative 4th hour
  From patients undergoing major abdominal surgery, a blood sample will be taken at Postop 4th Hour for serum NGAL analysis
Renal Doppler Resistive Index | Postoperative 4th hour
  Renal Doppler Resistive Index will be measured at the 4th hour after major abdominal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan OZYURT, Assoc. Prof., Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zeng X, McMahon GM, Brunelli SM, Bates DW, Waikar SS. Incidence, outcomes, and comparisons across definitions of AKI in hospitalized individuals. Clin J Am Soc Nephrol. 2014 Jan;9(1):12-20. doi: 10.2215/CJN.02730313. Epub 2013 Oct 31. PMID 24178971
- [Background] Muthukrishnan K, Parida S, Barathi SD, Badhe AS, Mishra SK. Doppler resistive index to reflect risk of acute kidney injury after major abdominal surgery: A prospective observational trial. Indian J Anaesth. 2019 Jul;63(7):551-557. doi: 10.4103/ija.IJA_189_19. PMID 31391618